CLINICAL TRIAL: NCT02681432
Title: Hyperthermic Intraperitoneal Chemotherapy With Paclitaxel for the Treatment of Patients With Recurrent or Primary Advanced Ovarian Cancer : A Randomised Phase 3 Study
Brief Title: Hyperthermic Intraperitoneal Chemotherapy With Paclitaxel in Advanced Ovarian Cancer
Acronym: hipecova
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PEDRO VILLAREJO CAMPOS (Other)
Collaborators: Hospital General de Ciudad Real (Other); University of Castilla-La Mancha (Other)
Responsible Party: Sponsor-Investigator, PEDRO VILLAREJO CAMPOS, MD, PhD.Associate Professor of Surgery. University of Castilla-La Mancha, Hospital General de Ciudad Real
Organization: Hospital General de Ciudad Real (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGCRCIRU001
Record Dates: First submitted 2016-01-25; First posted 2016-02-12 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Epithelial Ovarian Cancer
Keywords: HIPEC; ovarian cancer; peritoneal carcinomatosis
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms; Peritoneal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIPEC (Experimental): Primary ovarian cancer FIGO stage II, III or IV or recurrent
  Interventions: Drug: HIPEC
- No HIPEC (Active Comparator): Primary ovarian cancer FIGO stage II, III or IV or recurrent
  Interventions: Procedure: No HIPEC

INTERVENTIONS:
Drug: HIPEC — Cytoreductive surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) with Paclitaxel (175 mg/m2) for 60 minutes at 42-43 degrees.
  Arms: HIPEC
Procedure: No HIPEC — Cytoreductive surgery without HIPEC
  Arms: No HIPEC

SUMMARY:
Randomized clinical trial to asses the efficacy of closed abdomen hyperthermia intraperitoneal chemotherapy with paclitaxel in ovarian cancer.

DETAILED DESCRIPTION:
Randomized clinical trial performed in woman with epithelial primary ovarian cancer (stage FIGO II, III and IV) or tumor recurrence. A cytoreductive surgery will be perform in all of the patients include in the trial, and it will be assign at randomization:

* HIPEC-arm: cytoreductive surgery and hyperthermic intraperitoneal chemotherapy with paclitaxel (175 mg / m2) for 60 minutes at a temperature of 42-43º degrees; followed by postoperative systemic IV chemotherapy with carboplatin (AUC=6) and paclitaxel (175 mg/m2) for 6 cycles.
* No HIPEC-arm: Cytoreductive surgery followed by postoperative systemic IV chemotherapy with carboplatin (AUC=6) and paclitaxel (175 mg/m2) for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed epithelial ovarian cancer (stage II / III / IV disease of FIGO) or tumor recurrences (the women of childbearing age need to have a negative pregnancy test)
* Complete cytoreduction: Index CC0/CC1 cytoreduction (residual tumor size after surgery, no visible (CC0) or less than 0.25 cm (CC1))
* No extra-abdominal tumor disease
* Absence of heart failure. Adequate renal and hepatic functions
* Eastern Cooperative Oncology Group performance status 0-2 or Karnofsky performance status ≥ 70%

Exclusion Criteria:

* Patients with unresectable tumor or incomplete cytoreduction.
* Contraindications for treatment with paclitaxel: patients with severe hypersensitivity to paclitaxel or any of the excipients,pregnancy or lactation and patients with baseline neutrophil count <1.500/mm3 (<1.000/mm3 for patients with Kaposi sarcoma). Paclitaxel is also contraindicated in patients who have concurrent and severe infections.
* Extra-abdominal metastases or unresectable liver metastases
* Presence of other malignant tumor disease.
* Multisegmental complete bowel obstruction.
* Patients with severe medical problems that will preclude compliance with the study or with an unacceptable risk
* Patients who refuse treatment or consent to participate in study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | every 6 months till 36 months
  From the date of surgery to the date of death or to the end of study (follow up every 6 months till 3 years)

SECONDARY OUTCOMES:
Progression free survival | follow up every 6 months till 18 months
  From the date of surgery to the date of recurrence or to the end of study (follow up every 6 months till 18 months)

OTHER OUTCOMES:
Post-operative complications | adverse events within 30 days postoperatively (according to NCI criteria, Common Terminology Criteria for AE (CTCAE))
  Compare adverse events between study arms

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Villarejo Campos, MD, PhD, Principal Investigator — SESCAM
Locations (1):
- Hospital General Ciudad Real, Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munoz-Casares FC, Rufian S, Rubio MJ, Diaz CJ, Diaz R, Casado A, Arjona A, Munoz-Villanueva MC, Muntane J. The role of hyperthermic intraoperative intraperitoneal chemotherapy (HIPEC) in the treatment of peritoneal carcinomatosis in recurrent ovarian cancer. Clin Transl Oncol. 2009 Nov;11(11):753-9. doi: 10.1007/s12094-009-0438-3. PMID 19917539
- [Background] Jaaback K, Johnson N, Lawrie TA. Intraperitoneal chemotherapy for the initial management of primary epithelial ovarian cancer. Cochrane Database Syst Rev. 2016 Jan 12;2016(1):CD005340. doi: 10.1002/14651858.CD005340.pub4. PMID 26755441
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Background] Chua TC, Robertson G, Liauw W, Farrell R, Yan TD, Morris DL. Intraoperative hyperthermic intraperitoneal chemotherapy after cytoreductive surgery in ovarian cancer peritoneal carcinomatosis: systematic review of current results. J Cancer Res Clin Oncol. 2009 Dec;135(12):1637-45. doi: 10.1007/s00432-009-0667-4. Epub 2009 Aug 23. PMID 19701772
- [Background] Bijelic L, Jonson A, Sugarbaker PH. Systematic review of cytoreductive surgery and heated intraoperative intraperitoneal chemotherapy for treatment of peritoneal carcinomatosis in primary and recurrent ovarian cancer. Ann Oncol. 2007 Dec;18(12):1943-50. doi: 10.1093/annonc/mdm137. Epub 2007 May 11. PMID 17496308
- [Background] Kim JH, Lee JM, Ryu KS, Lee YS, Park YG, Hur SY, Lee KH, Lee SH, Kim SJ. Consolidation hyperthermic intraperitoneal chemotherapy using paclitaxel in patients with epithelial ovarian cancer. J Surg Oncol. 2010 Feb 1;101(2):149-55. doi: 10.1002/jso.21448. PMID 20035540
- [Background] Benedetti Panici P, Palaia I, Graziano M, Bellati F, Manci N, Angioli R. Intraperitoneal paclitaxel as consolidation treatment in ovarian cancer patients: a case control study. Oncology. 2010;78(1):20-5. doi: 10.1159/000287968. Epub 2010 Feb 24. PMID 20185937
- [Background] de Bree E, Rosing H, Filis D, Romanos J, Melisssourgaki M, Daskalakis M, Pilatou M, Sanidas E, Taflampas P, Kalbakis K, Beijnen JH, Tsiftsis DD. Cytoreductive surgery and intraoperative hyperthermic intraperitoneal chemotherapy with paclitaxel: a clinical and pharmacokinetic study. Ann Surg Oncol. 2008 Apr;15(4):1183-92. doi: 10.1245/s10434-007-9792-y. Epub 2008 Feb 1. PMID 18239973
- [Background] Seretis C, Youssef H. Quality of life after cytoreductive surgery and intraoperative hyperthermic intraperitoneal chemotherapy for peritoneal surface malignancies: a systematic review. Eur J Surg Oncol. 2014 Dec;40(12):1605-13. doi: 10.1016/j.ejso.2014.08.477. Epub 2014 Sep 6. PMID 25242382